CLINICAL TRIAL: NCT05526820
Title: A Randomized, Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Live Attenuated Varicella Vaccine Combined With Inactivated Hepatitis A Vaccine
Brief Title: A Study of Combined Immunization With Live Attenuated Varicella Vaccine and Inactivated Hepatitis A Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VZV-4001
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combined immunization group (Experimental): 225 participants received one dose of live attenuated varicella vaccine and the first dose inactivated hepatitis A vaccine on day 0 and the second dose of inactivated hepatitis A vaccine on day 180.
  Interventions: Biological: The live attenuated varicella vaccine and the inactivated hepatitis A vaccine
- The Non-combined immunization group (Active Comparator): 225 participants received one dose of live attenuated varicella vaccine on day 0,the first dose of inactivated hepatitis A vaccine on day 42 and the second dose of inactivated hepatitis A vaccine on day 222.
  Interventions: Biological: The live attenuated varicella vaccine and the inactivated hepatitis A vaccine

INTERVENTIONS:
Biological: The live attenuated varicella vaccine and the inactivated hepatitis A vaccine — The live attenuated varicella vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd,the inactivated hepatitis A vaccine was manufactured by Sinovac Biotech Co., Ltd.
  The live attenuated varicella vaccine:live varicella-zoster virus in 0.5 mL of sucrose, sodium glutamate,sodium chloride,potassium chloride,sodium dihydrogen phosphate, potassium dihydrogen phosphate and injection water per injection.
  The inactivated hepatitis A vaccine:250 U inactivated virus in 0.5mL of aluminium hydroxide solution per injection.
  All subjects received hepatitis A vaccine in the upper left arm and varicella vaccine in the upper right arm.

SUMMARY:
This study is a randomized and controlled Phase IV clinical trial.The purpose of this study is to evaluate the immunogenicity and safety of combined immunization with live attenuated varicella vaccine and inactivated hepatitis A vaccine in children aged 12-15 months.

DETAILED DESCRIPTION:
This study is a randomized and controlled phase IV clinical trial in children aged 1 year old (12-15 months).The purpose of this study is to evaluate the immunogenicity and safety of live attenuated varicella vaccine co-administration with inactivated hepatitis A vaccine .The live attenuated varicella vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd,the inactivated hepatitis A vaccine was manufactured by Sinovac Biotech Co., Ltd.A total of 450 subjects aged 1 year old (12-15 months) were be enrolled.Subjects were be randomly divided into 2 groups in a ratio of 1:1.Subjects in the combined immunization group received one dose of live attenuated varicella vaccine and the first dose inactivated hepatitis A vaccine on day 0 and the second dose of inactivated hepatitis A vaccine on day 180.Subjects in the Non-combined immunization group received one dose of live attenuated varicella vaccine on day 0,the first dose of inactivated hepatitis A vaccine on day 42 and the second dose of inactivated hepatitis A vaccine on day 222.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child aged 1 year old (12-15 months old);
* Proven legal identity;
* The subjects'guardians should be capable of understanding the informed consent form, and such form should be signed prior to enrolment.

Exclusion Criteria:

* History of vaccination of varicella vaccine or hepatitis A vaccine.
* Previous history of varicella infection or hepatitis A infection;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Thyroid disease or history of thyroidectomy, asplenia,functional asplenia,asplenia or splenectomy resulting from any condition;
* Suffering from serious chronic diseases, serious cardiovascular diseases, liver and kidney diseases, malignant tumors, etc;
* Family history of psychosis,severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) within 6 months before enrollment;
* Receipt of blood products within the past 3 months;
* Receipt of other investigational vaccines or drugs within 28 days prior to receiving the investigational vaccine;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Armpit temperature in subjects with fever prior to vaccination with the investigational vaccine. 37.4 ℃;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of the varicella antibody | 42 days after immunization of live attenuated varicella vaccine
  Seroconversion rate of varicella antibody 42 days after immunization of live attenuated varicella vaccine.
Seroconversion rates of anti-HAV antibody | 30 days after full immunization with hepatitis A vaccine
  Seroconversion rate of anti-HAV antibody 30 days after full immunization with hepatitis A vaccine.

SECONDARY OUTCOMES:
Seropositive rates of varicella antibody | 42 days after immunization of live attenuated varicella vaccine
  Seropositive rates of varicella antibody 42 days after immunization of live attenuated varicella vaccine.
GMT of varicella antibody | 42 days after immunization of live attenuated varicella vaccine
  GMT of varicella antibody 42 days after immunization of live attenuated varicella vaccine.
GMI of varicella antibody | 42 days after immunization of live attenuated varicella vaccine
  GMI of varicella antibody 42 days after immunization of live attenuated varicella vaccine.
Seropositive rates of anti-HAV antibody | 30 days after full immunization with hepatitis A vaccine
  Seropositive rates of anti-HAV antibody 30 days after full immunization with hepatitis A vaccine.
GMC of anti-HAV antibody | 30 days after full immunization with hepatitis A vaccine
  GMC of anti-HAV antibody 30 days after full immunization with hepatitis A vaccine.
GMI of anti-HAV antibody | 30 days after full immunization with hepatitis A vaccine
  GMI of anti-HAV antibody 30 days after full immunization with hepatitis A vaccine.
The incidence of adverse events | within 0-42 days (or 0-30 days) after each dose of vaccine
  Incidence of adverse events within 0-42 days (or 0-30 days) after each dose of vaccine.
The incidence of local and systemic solicitation adverse reactions | Within 0-14 days (or 0-7 days) after each dose of vaccine
  The incidence of local and systemic solicitation adverse reactions within 0-14 days (or 0-7 days) after each dose of vaccine.
The incidence of serious adverse events (SAE) | Within 42 days (or 30 days) after administration of each dose of vaccine
  The incidence of serious adverse events (SAE) within 42 days (or 30 days) after administration of each dose of vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Dianmin Kang, Principal Investigator — Shandong Provincial Center for Disease Prevention and Control
Locations (1):
- Feicheng Center for Disease Control and Prevention, Tai’an, Shandong, China

REFERENCES:
- [Derived] Sun D, Yu D, Du Z, Jia N, Liu X, Sun J, Xu Q, Sun Z, Luan C, Lv J, Xiong P, Zhang L, Sha X, Gao Y, Kang D. Immunogenicity and safety of a live attenuated varicella vaccine co-administered with inactive hepatitis A vaccine: A phase 4, single-center, randomized, controlled trial. Hum Vaccin Immunother. 2023 Dec 31;19(1):2161789. doi: 10.1080/21645515.2022.2161789. Epub 2023 Jan 2. PMID 36593652